CLINICAL TRIAL: NCT01745653
Title: Monocentric, Randomized, Single Blinded Study Designed to Evaluate the Effect of Low Level Laser Therapy on Pain Occurring After Insertion of an Orthodontic Device : the "Quadhelix"
Brief Title: Effect of Low Level Laser Therapy on Pain Occurring After Insertion of an Orthodontic Device
Acronym: Ortholaser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRD11/3-J
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Bad Molar Teeth Arrangement Requiring Orthodontic Device
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low level laser therapy (Experimental): Low level laser (970nm) will be delivered on the mucous membrane in regard to the first molar teeth on which rings of the quadhelix have been settled.
  Interventions: Device: Low level laser therapy
- sham procedure (Sham Comparator): Same procedure than experimental arm except that the laser is not activated.
  Interventions: Procedure: sham procedure
- no intervention (No Intervention): no intervention : Patient received the quadhelix with nothing else

INTERVENTIONS:
Device: Low level laser therapy
  Other Names: low level laser therapy (970nm) (SIROLaser advance material of SIRONA dental systems laboratory)
  Arms: Low level laser therapy
Procedure: sham procedure
  Other Names: Same intervention than experimental arm except that the laser is not activated
  Arms: sham procedure

SUMMARY:
Thus study consists of evaluating the effect of low level therapy on pain induced by insertion of an orthodontic device (the "quadhelix"). Each day during the first seven days post procedure, the level of pain will be reported on an analogic visual scale.

As secondary objectives, intake of antalgics and type of swallowed food (soft or tough) will also be daily registered.

DETAILED DESCRIPTION:
Patient will be randomized into one of the 3 following arms :

* arm 1 (experimental) : administration of Low Level Laser Therapy just after insertion of the quadhelix.
* arm 2 (sham procedure) : material necessary to perform Low Level Laser Therapy will be installed but the laser will not be activated.
* arm 3 (no intervention): material necessary to perform Low Level Laser Therapy will NOT be installed

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 15 years old who need to receive an orthodontic device ("quadhelix)
* informed consent form signed by parents who should be affiliated to French health insurance (french Social security)

Exclusion Criteria:

* malignant facial tumor
* not able to read or write correctly and thus not able to complete the questionnaire
* allergic or intolerant to paracetamol
* Informed consent not obtained

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of low level laser therapy on pain induced by insertion of the quadhelix (orthodontic device) | change from baseline pain at 7 days
  Each day during the first week post procedure, patient will record intensity of his/her pain on an analogic visual scale

SECONDARY OUTCOMES:
effect of low level laser therapy on intake of antalgics | change from baseline antalgics intake at 7 days
  Each day during the first week post procedure, patient will record his/her intake of antalgics
quality of food intake | change from baseline quality of food intake at 7 days
  Each day during the first week post procedure, patient will answer (on a questionnaire) to questions concerning his/her intake of food (type of food (soft or not)).

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Universitary Hospital, Nantes, Loire Atlantique, France